CLINICAL TRIAL: NCT05288699
Title: Brief Personalized Feedback Intervention for Latinx Hazardous Drinkers: A Community-Based Intervention
Brief Title: Mobile App for Latinx Hazardous Drinkers With Clinical Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael J. Zvolensky, Ph.D. (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Michael J. Zvolensky, Ph.D., Distinguished Professor, University of Houston
Organization: University of Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003577
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Abuse; Anxiety
Keywords: Latinx; Hispanic; Personalized Feedback Intervention
MeSH Terms: conditions — Alcoholism; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aliento (Experimental): Participants complete the brief (~30 minute) intervention at baseline and will have access to intervention material for up to 3-months after the baseline appointment via the mobile health application.
  Interventions: Behavioral: Aliento

INTERVENTIONS:
Behavioral: Aliento — Aliento is a culturally adapted, brief, personalized feedback intervention (PFI) to address alcohol misuse in the context of clinical anxiety delivered via a mobile application.

SUMMARY:
The purpose of this study is to develop and examine a culturally adapted, brief, integrated, Spanish language mobile health application for the Android platform, optimized to deliver a personalized feedback intervention (PFI) designed to enhance knowledge regarding adverse anxiety-alcohol interrelations, increase motivation and intention to reduce hazardous drinking, and reduce positive attitudes and intention regarding anxiety-related alcohol use among Latinx hazardous drinkers with clinical anxiety.

DETAILED DESCRIPTION:
Investigators will develop a culturally adapted, brief, single-session, Spanish language, PFI delivered via a mobile health application for the Android platform through an iterative approach using expert input and focus groups. Next, Latinx hazardous drinkers with clinical anxiety will assess program navigation and conduct usability testing. Finally, Latinx hazardous drinkers with clinical anxiety will be recruited to complete the final prototype of the mobile health application in order to evaluate the feasibility, acceptability, and initial effects. Initial screening will be conducted via telephone; baseline and post-treatment data will be collected in-person; and 1-week, 1-month, and 3-months follow-up data will be collected remotely.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* self-identified as Latinx or Hispanic
* fluent in Spanish
* current hazardous drinking pattern
* current clinical anxiety
* able to provide written, informed consent
* owning an Android smartphone

Exclusion Criteria:

* currently involved in alcohol or other substance use program
* concurrent use of medication for anxiety or depression
* current engagement in psychotherapy for anxiety or depression

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test | Change from Baseline Pre PFI Completion to 3-months Post PFI Completion
  The Alcohol Use Disorders Identification Test will be used to assess drinking quantity, craving, and related consequences to alcohol use. The 10 items are rated with various Likert-type scales. The measure produces a total score by adding all of the items of the measure with higher scores indicating greater problems with alcohol (possible range 0 to 40).
Overall Anxiety Severity and Impairment Scale | Change from Baseline Pre PFI Completion to 3-months Post PFI Completion
  The 5-item Overall Anxiety Severity and Impairment Scale will be used to assess anxiety symptom severity and impairment. Each of the items is rated on a Likert-type scale ranging from 0 to 4. Items are summed to produce a total score (possible range 0 to 20).

SECONDARY OUTCOMES:
Motivation to Reduce Alcohol Consumption Scale | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The 1-item Motivation to Reduce Alcohol Consumption Scale will be used to measure current motivation/intention to reduce alcohol. Participants will be asked to select the statement that best describes their motivation/intention to reduce drinking (e.g., "I really want to cut down on drinking alcohol and intend to in the next month"). Higher scores on this measure indicate greater motivation/intention to reduce alcohol consumption (possible range (0-7).
Modified Drinking Motives Questionnaire-Revised | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The Modified Drinking Motives Questionnaire-Revised will be used to assess expectancies of drinking. For the current study, the 4-item "Coping-anxiety" subscale will be used as a measure of expectancies of drinking to reduce/cope with anxiety. The measure utilizes a 5-point Likert scale ranging from 1 (almost never/never) to 5 (almost always/always). Scores are averaged with higher scores indicating greater expectancies of drinking to reduce/cope with anxiety (possible range 1 to 5).
Alcohol Attitudes Scale | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The 7-item Alcohol Attitudes Scale will be utilized to measure maladaptive attitudes for drinking (e.g., "Drinking alcohol is good"). Items are rated on a Likert-type scale from 1 (strongly disagree) to 7 (strongly agree). Scores will be averaged to create a composite score (possible range 1 to 7). Higher scores indicate greater maladaptive attitudes for drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Principal Investigator — University of Houston
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Treatment Outcomes, and Racial Equity, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.